CLINICAL TRIAL: NCT06184477
Title: Pediatric Tonsillectomy: Surgical Experience And Prolonged Hospitalization
Brief Title: The Relationship Between Prolonged Hospitalization and Surgical Experience in Pediatric Tonsillectomy Cases.
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fazıl Necdet Ardıç, Prof Dr, Pamukkale University
Other Study IDs: 15
Record Dates: First submitted 2023-12-09; First posted 2023-12-28 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Sleep Apnea; Tonsillitis Recurrent
Keywords: Tonsillectomy; Prolonged hospitalization
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prolonged hospitalization after tonsillectomy: Prolonged hospitalization refers to prolonged discharge time and readmission.
  Interventions: Other: PEDIATRIC TONSILLECTOMY; SURGICAL EXPERIENCE AND PROLONGED HOSPITALIZATION
- normal hospitalization time: normal hospitalization time for pediatric patients accepted as 1 night stay.
  Interventions: Other: PEDIATRIC TONSILLECTOMY; SURGICAL EXPERIENCE AND PROLONGED HOSPITALIZATION

INTERVENTIONS:
Other: PEDIATRIC TONSILLECTOMY; SURGICAL EXPERIENCE AND PROLONGED HOSPITALIZATION — we aim to compare hospitalization times of pediatric patients that operated by expert surgeon or young surgeon

SUMMARY:
Guided by the expertise of a seasoned surgeon at the tertiary care hospital, the training program includes performing tonsillectomy starting from the 6th month. The clinical protocol at the hospital dictates a standard one-night hospital stay for all patients, but there is potential to extend the duration in specific cases. The study endeavors to explore the correlation between extended hospitalization, surgical proficiency, patient-specific factors, and postoperative complications in pediatric patients who underwent tonsillectomy and/or adenotonsillectomy at the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 18 years of age having tonsillectomy surgery
* Patients whose records are available in the hospital archive

Exclusion Criteria:

* Inadequate information in files

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A retrospective analysis was conducted on tonsillectomy patients under the age of 18, who underwent surgery at our clinic between 2019 and 2023.
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Incidence of hospitalization lasting more than 24 hours | december'23- january'24

SECONDARY OUTCOMES:
Incidence of postoperative complications | december'23- january'24
  incidence of bleeding, respiratory problems

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No